CLINICAL TRIAL: NCT01470287
Title: A Phase-III, Single Arm, Multi-Center, Open-Label Study to Assess the Immunogenicity, Safety and Tolerability of a Fully Liquid Pentavalent Vaccine (DTwP-Hib-HepB Vaccine) When Administered to Indian Infants at 6, 10, and 14 Weeks of Age
Brief Title: Immunogenicity, Safety and Tolerability of a Fully Liquid Pentavalent (DTwP-Hib-Hep B) Vaccine in Infants 6-8 Weeks of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V66_05
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Hemophilus Influenzae B
Keywords: Infants,; Immunogenicity,; Safety
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B | interventions — DtwP-HepB-Hib vaccine

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: DTwP-HepB-Hib Vaccine

INTERVENTIONS:
Biological: DTwP-HepB-Hib Vaccine — Open label, Single arm study to evaluate immunogenicity, safety and tolerability of a fully liquid pentavalent (DTwP-HepB-Hib) vaccine in infants of 6-8 weeks of age.

SUMMARY:
This study will evaluate immunogenicity, safety and tolerability of fully liquid pentavalent vaccine (DTwP-Hib-HepB Vaccine) in infants 6-8 weeks of age.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥ 42 days to ≤ 64 days of age.
2. Written informed consent obtained from either parents/ legal guardian after the nature of the study has been explained according to local regulatory requirements

Exclusion Criteria:

1. Subjects whose parents or legal guardians are unwilling or unable to give written informed consent to participate in the study.
2. History of previous immunization with a vaccine containing any of the 5 antigen components of investigational vaccine.
3. History of anaphylactic shock(immediate hypersensitivity reactions), urticaria or other allergic reactions after previous vaccination or known hypersensitivity to any vaccine component.
4. Administration of parenteral immunoglobulin preparation and/or blood products since birth.

Ages: 42 Days to 64 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Seroprotection rate one month after the last dose of vaccine administration | One month after last vaccination

SECONDARY OUTCOMES:
Seroprotection rate and GMCs one month after the last vaccine administration | One month after last vaccination

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Rajarajeshwari Medical College and Hospital, Bangalore, Karnataka
  - Bharathi Vidyapeeth University, Pune, Maharashtra
  - Medical College Kolkata, Kolkata, West Bengal

REFERENCES:
- [Derived] Eregowda A, Lalwani S, Chatterjee S, Vakil H, Ahmed K, Costantini M, Lattanzi M. A phase III single arm, multicenter, open-label study to assess the immunogenicity and tolerability of a pentavalent DTwP-HepB-Hib vaccine in indian infants. Hum Vaccin Immunother. 2013 Sep;9(9):1903-9. doi: 10.4161/hv.25166. Epub 2013 Jun 19. PMID 23783081